CLINICAL TRIAL: NCT06784934
Title: Mindful Minds: Acceptability and Feasibility of Mindfulness-Based Neurofeedback Training for Racial and Ethnic Minority Scholars
Brief Title: Mindful Minds: Mindfulness-Based Neurofeedback for Underrepresented College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amelia Saul, PhD, CTRS, BCB, Assistant Teaching Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 800-020-774; U54MD012393 (NIH)
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-02

CONDITIONS: Academic Performance; Anxiety
Keywords: neurofeedback; underrepresented population; college students; academic performance; anxiety; mindfulness meditation; wearable devices; biofeedback; Heart Rate Variability; Alpha Neurofeedback
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Neurofeedback (Experimental): For the experimental group, participants will engage in a mindfulness-based neurofeedback training protocol designed to enhance academic performance and reduce performance anxiety. The intervention involves the use of NeuroSky and BrainTrain technology to provide real-time feedback on brain activity, helping participants develop better self-regulation skills. The training incorporates guided mindfulness exercises focused on promoting relaxation and sustained attention.
  After the training with the researcher, the experimental group participants will go home and practice independently (10 -15 minutes of mindfulness-based neurofeedback training once daily) with weekly 10-minute virtual check-ins for 4 weeks. Participants will also be asked to record 5 minutes of heart rate variability (HRV) data using the OptimalHRV device twice a day to measure their HRV. At the end of the study, participants will return to the lab for one final mindfulness-meditation session.
  Interventions: Device: NeuroSky Mindfulness-Based Neurofeedback
- Business as Usual (No Intervention): The control group participants will not engage in mindfulness-based neurofeedback training. Participants in the control group will continue their daily routines without meditation for 4 weeks. Heart rate variability (HRV) will be monitored using the OptimalHRV device to monitor HRV, but no intervention will be provided. Weekly 10-minute virtual check-ins with the research team will ensure compliance, address questions, and maintain engagement. Data collected from the OptimalHRV device will provide a baseline for comparison, helping to evaluate the effectiveness of the neurofeedback intervention in the experimental group.

INTERVENTIONS:
Device: NeuroSky Mindfulness-Based Neurofeedback — NeuroSky will monitor participants' brain response to the intervention and provide feedback based on the participants' performance. Neurofeedback Intervention: When practicing the mindfulness-based intervention, NeuroSky will provide instructions before beginning the sessions. Dr. Saul will assist with set up and answer any questions. The apps audio and visual feedback will assist the participants as they practice mindfulness meditation. Participants in the experimental group will practice for 10 minutes in the lab during Sessions 1 and 5 and then at home for 10-20 minutes daily for 4 weeks with weekly 10-minute virtual check-ins with Dr. Saul to ensure acceptability and feasibility. Dr. Saul will also monitor participants' progress using the secure participant portal and de-identified usernames available through NeuroSky.
  Arms: Mindfulness Neurofeedback

SUMMARY:
The study examines the efficacy of a mindfulness-based neurofeedback protocol designed to improve academic performance and reduce performance anxiety in racial and ethnic minority college students. Using NeuroSky and BrainTrain technology, the intervention incorporates mindfulness principles to enhance participants' self-regulation skills. Continuous heart rate variability (HRV) data is collected to assess stress levels, sleep, and exercise. The research aims to explore the acceptability and feasibility of this approach, with the goal of addressing academic performance and anxiety in this population.

DETAILED DESCRIPTION:
The United States has witnessed a notable increase in the enrollment of racial and ethnic minority students (i.e., "The minority racial and ethnic groups defined by Office of Management and Budget's (OMB) are American Indian or Alaska Native, Asian, Black or African American, and Native Hawaiian or Pacific Islander. The ethnicity used is Latino or Hispanic"). With the rise in college enrollment has also come concerns about the challenges racial and ethnic minority students are facing, such as "experiencing microaggressions, discrimination, imposter syndrome, and negative campus climate," which have been found to contribute to mental health problems for minority college students. Those who identify as more than one race had the highest rate of anxiety (39.8%), followed by American Indian/Alaskan Native (39.1%), Arab/Arab American (35.2%) and Latino (35.2%).6 However, the majority of research about college students' mental health status and treatment is focused on the general college student population, with extensive studies having only small subsets of racial and ethnic minority student representation. Given the ubiquity of mental health challenges in college students, the development of an easily utilized, readily available, inexpensive, with minimal side-effects intervention is needed. Neurofeedback and mindfulness have both been found to show significant improvements in performance enhancement, anxiety reduction, and improved focus/awareness. Through continuous neurofeedback interventions, individuals tend to improve interoceptive awareness and develop mechanisms to facilitate emotional control. Mindfulness meditation can help individuals gain control of their attention, which may, in turn, help to facilitate control of thoughts and emotions. Currently, there is little research on the benefits of neurofeedback using mindfulness-based interventions to improve academic performance in students from racial and ethnic minority backgrounds. This research program responds to the urgent need for targeted interventions to enhance academic success and improve mental health among racial and ethnic minority students in higher education. Using a randomized control trial, 36 participants will be randomly assigned to either the 4-week mindfulness-based neurofeedback intervention or business as usual. The investigators hypothesize that participants in the experimental group will significantly improve test performance and reduce academic anxiety compared to the control group. Focused on examining the acceptability and feasibility of a mindfulness-based neurofeedback intervention, the study aims to address performance anxiety and improve test performance as well as mental health by providing real-time feedback and objective analysis to overcome the limitations of traditional stress management programs. The research also aims to offer a more accessible and practical approach, contributing valuable insights to promote equitable outcomes for underrepresented students.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years old
* Currently enrolled in a 4-year university
* Individuals from an ethnic or racial minority background (i.e., "The minority racial and ethnic groups defined by Office of Management and Budget's (OMB) are American Indian or Alaska Native, Asian, Black or African American, and Native Hawaiian or Pacific Islander. The ethnicity used is Latino or Hispanic.")

Exclusion Criteria:

* Severe depression (cut off score of 15 or higher on Patient Health Questionnaire 9 (PHQ-9))
* Previously receiving biofeedback training.
* Severe medical condition (e.g., pacemaker, cardiac arrhythmia, hypertension, diabetes).
* Showing symptoms of psychosis
* Having a neurological condition (e.g., Parkinson's disease) that would complicate the interpretation of physiological data.
* Taking medications such as SSRIs, alpha/beta-blockers, or withdrawal or maintenance medications (e.g., Librium, methadone)
* Using substances such as tobacco and illicit drugs, and 8)alcohol consumption as defined by National Institute of Health (NIH) as "more than 2 drinks (1 drink for women) in a day or drinking more than 5 drinks (4 for women) on the same occasion (i.e., at the same time or within a couple of hours of each other) on at least 1 day in the past month" are excluded due to their potential to affect the data.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Academic Performance | From enrollment to the end of treatment at 4 weeks
  Trier Social Stress Test will be utilized to induce performance anxiety through a mock job interview and mental arithmetic task conducted in front of a non-responsive committee. This test uses a standardized protocol that not only facilitates a more robust evaluation of our intervention but also elevates the ecological validity of the study by assessing its effects in a real-life scenario. The social stress test not only facilitates a more robust evaluation of our intervention but also elevates the ecological validity of the study by assessing its effects in a real-life scenario.
Academic Anxiety with Academic Anxiety Scale | From enrollment to the end of treatment at 4 weeks
  The Academic Anxiety Scale (AAS) will be used to examine performance anxiety (Aim 1). This 11-item questionnaire uses a 4-point Likert Scale (1 = not at all typical of me to 4 = very typical of me) and measures broader aspects of academic-based anxiety beyond cognitive factors. The AAS includes items designed to assess apprehension and anxiety in academic settings, with high reliability (split-half Guttman reliability of 0.91 and Cronbach's Alpha of 0.94).
Acceptability | From enrollment to the end of treatment at 4 weeks
  Semi-structured interviews will be conducted during the weekly check-ins to further our understanding of the intervention's acceptability utilizing qualitative techniques such as thematic analysis.
Academic Anxiety with Beck Anxiety Inventory | From enrollment to the end of treatment at 4 weeks
  The Beck Anxiety Inventory (BAI) will measure generalized anxiety using a 21-item Likert scale (0 to 3) to assess how distressing anxiety symptoms have been over the past week. Scores range from 0 to 63, with levels categorized as minimal (0-7), mild (8-15), moderate (16-25), and severe (30-63). The BAI has been widely used among racially diverse groups. The investigators hypothesize that BAI scores will vary significantly from pre- to post-intervention.
Feasibility | From enrollment to the end of treatment at 4 weeks
  Semi-structured interviews will be conducted during the weekly check-ins to further our understanding of the intervention's feasibility utilizing qualitative techniques such as thematic analysis.

SECONDARY OUTCOMES:
Attention with Integrated Visual and Auditory Continuous Performance Test | From enrollment to the end of treatment at 4 weeks
  The Integrated Visual and Auditory Continuous Performance Test (IVA-2) will be used to assess attention as a secondary outcome. This computerized test measures both visual and auditory attention, providing an overall score of attentional functioning and response control. It evaluates sustained attention, impulsivity, and processing speed through a series of tasks requiring quick and accurate responses.The scores range from 0 to 145, with a mean of 100 and a standard deviation of 15. Higher scores reflect better performance. Scores of zero are valid, indicating performance 6.65 SD below average. The test includes a validity check (p < .01) for random responses, allowing scores to be set to zero if effort was made. Rating scales are available for additional validity assessment.
Increased Alpha Activity | From enrollment to the end of treatment at 4 weeks
  The NeuroSky device will be used to measure alpha brainwave activity, a marker of relaxation and focused attention, as a secondary outcome. Mindfulness-based neurofeedback training will aim to enhance alpha activity by providing participants with real-time feedback on their brainwave patterns. During each session, participants will learn to modulate their alpha levels through mindfulness techniques, fostering a state of calm alertness. Increased alpha activity is associated with improved emotional regulation, reduced stress, and enhanced cognitive functioning. Pre- and post-intervention alpha activity levels will be compared to evaluate the effectiveness of the mindfulness-based neurofeedback training.
Attention with Mental Stress Assessment | From enrollment to the end of treatment at 4 weeks
  The Mental Stress Assessment (MeSA) will also assess attention by measuring physiological responses during tasks designed to induce and evaluate stress-related attentional shifts.
Heart Rate Variability | From enrollment to the end of treatment at 4 weeks
  Heart Rate Variability (HRV) will be measured using the OptimalHRV device. We will examine HRV to determine if participants HRV increased from pre- to post-test which would be an indication of improved autonomic nervous system balance.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia D Saul, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators recognize the importance of sharing Individual Participant Data (IPD) to advance scientific discovery and promote transparency in research. While protecting participant privacy and adhering to ethical and regulatory guidelines remains a top priority, the investigators are exploring options to make IPD from this study available under appropriate conditions. Any shared data will be fully de-identified to safeguard participant privacy and minimize the risk of re-identification. Data sharing will occur through secure, controlled-access repositories or upon request, with approval contingent on a data use agreement to ensure responsible use. Furthermore, data sharing will align with the informed consent provided by participants, respecting their rights and preferences. The investigators will also limit shared data to specific research purposes that align with the study's objectives and have the potential to benefit the broader scientific community.

REFERENCES:
- [Background] Rogers JM, Johnstone SJ, Aminov A, Donnelly J, Wilson PH. Test-retest reliability of a single-channel, wireless EEG system. Int J Psychophysiol. 2016 Aug;106:87-96. doi: 10.1016/j.ijpsycho.2016.06.006. Epub 2016 Jun 16. PMID 27318008
- [Background] Stinson B, Arthur D. A novel EEG for alpha brain state training, neurobiofeedback and behavior change. Complement Ther Clin Pract. 2013 Aug;19(3):114-8. doi: 10.1016/j.ctcp.2013.03.003. Epub 2013 Apr 19. PMID 23890456
- [Background] Hunkin H, King DL, Zajac IT. Evaluating the feasibility of a consumer-grade wearable EEG headband to aid assessment of state and trait mindfulness. J Clin Psychol. 2021 Nov;77(11):2559-2575. doi: 10.1002/jclp.23189. Epub 2021 Jun 1. PMID 34061998
- [Background] Hunt CA, Hoffman MA, Mohr JJ, Williams AL. Assessing Perceived Barriers to Meditation: the Determinants of Meditation Practice Inventory-Revised (DMPI-R). Mindfulness (N Y). 2020 May;11(5):1139-1149. doi: 10.1007/s12671-020-01308-7. Epub 2020 Feb 10. PMID 33664878
- [Background] Russell L, Orellana L, Ugalde A, Milne D, Krishnasamy M, Chambers R, Livingston PM. Exploring Knowledge, Attitudes, and Practice Associated With Meditation Among Patients With Melanoma. Integr Cancer Ther. 2018 Jun;17(2):237-247. doi: 10.1177/1534735417699514. Epub 2017 Mar 24. PMID 28627247
- [Background] Allen AP, Kennedy PJ, Dockray S, Cryan JF, Dinan TG, Clarke G. The Trier Social Stress Test: Principles and practice. Neurobiol Stress. 2016 Nov 12;6:113-126. doi: 10.1016/j.ynstr.2016.11.001. eCollection 2017 Feb. PMID 28229114
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Cassady JC, Pierson EE, Starling JM, editors. Predicting student depression with measures of general and academic anxieties. Frontiers in Education; 2019: Frontiers Media SA.
- [Background] Bigliassi M, Galano BM, Lima-Silva AE, Bertuzzi R. Effects of mindfulness on psychological and psychophysiological responses during self-paced walking. Psychophysiology. 2020 Apr;57(4):e13529. doi: 10.1111/psyp.13529. Epub 2020 Jan 17. PMID 31953844
- [Background] Saul AD, Fish MT. Anxiety and college students: The benefits of mindfulness-based meditation. Recreation, Parks, and Tourism in Public Health. 2019;3(1):139-54.
- [Background] Saul AD. The Efficacy of an Evidence-Based Biofeedback Intervention to Reduce Anxiety in College Students: East Carolina University; 2021.
- [Background] Fish MT, Saul AD. The gamification of meditation: a randomized-controlled study of a prescribed mobile mindfulness meditation application in reducing college students' depression. Simulation & Gaming. 2019;50(4):419-35.
- [Background] Russ SL, Maruyama G, Sease TB, Jellema S. Do early experiences matter? Development of an Early Meditation Hindrances Scale linked to novice meditators' intention to persist. Psychology of Consciousness: Theory, Research, and Practice. 2017;4(3):274.
- [Background] Kiken LG, Garland EL, Bluth K, Palsson OS, Gaylord SA. From a state to a trait: Trajectories of state mindfulness in meditation during intervention predict changes in trait mindfulness. Pers Individ Dif. 2015 Jul 1;81:41-46. doi: 10.1016/j.paid.2014.12.044. PMID 25914434
- [Background] Garland EL, Hanley A, Farb NA, Froeliger BE. State Mindfulness During Meditation Predicts Enhanced Cognitive Reappraisal. Mindfulness (N Y). 2015 Apr 1;6(2):234-242. doi: 10.1007/s12671-013-0250-6. PMID 26085851
- See also: IVA-2 Attention Assessment — https://www.braintrain.com/iva2/
- See also: MeSA Attention Assessment — https://www.braintrain.com/mesa/
- See also: Calm Awareness App — https://apps.apple.com/il/app/calm-awareness/id6450367887
- See also: BrainTrain SmartMind — https://www.braintrain.com/smartmind4-edu/